CLINICAL TRIAL: NCT07055984
Title: Predicting Outcomes in Posttransplant Diabetes Mellitus Via microRNA
Acronym: POD-MIR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Martin (Other)
Responsible Party: Principal Investigator, Matej Vnucak, Study coordinator, University Hospital, Martin
Other Study IDs: University hospital Martin
Record Dates: First submitted 2025-06-09; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus; Kidney Transplant
Keywords: post-transplant diabetes mellitus; microRNA; kidney transplantation
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients after primary kidney transplantation without type 1 or type 2 diabetes melltus

SUMMARY:
The study aims to improve the prediction and early detection of post-transplant diabetes mellitus (PTDM) in kidney transplant recipients. The investigators are investigating whether specific microRNA profiles measured 3 months after transplantation can reliably predict the development of PTDM within the following one to two years.

Additionally, the investigators are evaluating how traditional risk factors-such as age, immunosuppressive therapy, obesity, and infections like CMV-interact with these microRNA markers.

The ultimate goal of this research is to identify early indicators of blood sugar issues, enabling timely interventions to improve health outcomes and personalize patient care after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing kidney transplantation.
* Absence of pre-existing type 1 or type 2 diabetes mellitus.
* Willingness to provide informed consent and comply with study procedures.

Exclusion Criteria:

* Pre-existing type 1 or type 2 diabetes mellitus.
* Previous organ transplantation.
* Severe comorbidities that could confound the assessment of PTDM (e.g., pancreatic disease).
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: kidney transplant recipietns after pirmary kidney transplantation from post mortem or libing kidney donor.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2028-04-28 (Estimated); Study Completion 2029-04-28 (Estimated)

PRIMARY OUTCOMES:
To identify a panel of microRNAs at 3 months post-kidney transplant that are significantly associated with the development of PTDM within a defined follow-up period (e.g., 1 year, 2 years). | From enrollment to the end - 12 months
  This measure quantifies the count of miRNAs that show statistically significant differential expression between patients who develop PTDM and those who do not within the follow-up period. The significance is determined based on adjusted p-values (<0.05) and fold-change thresholds (e.g., >2 or <0.5). The data will be summarized as the total number of miRNAs passing these criteria for each patient group, providing a comparison of miRNA profiles at 3 months post-transplant.

CONTACTS AND LOCATIONS:
Locations (2):
- Slovakia (2):
  - Transplant-nephorlogy department, Martin
  - University hospital Martin, Martin

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT07055984/Prot_SAP_000.pdf